CLINICAL TRIAL: NCT05387317
Title: A Randomised Controlled Trial to Assess the Immunogenicity, Safety & Reactogenicity of Standard Dose Versus Fractional Doses of COVID-19 Vaccines (Pfizer-BioNTech, AstraZeneca or Moderna) Given as a Booster Dose After Priming With Coronavac or AstraZeneca in Healthy Adults in Indonesia
Brief Title: Evaluation of COVID-19 Vaccines Given as a Booster in Healthy Adults in Indonesia (MIACoV Indonesia)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial cancelled prior to commencement due to lack of funding.
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Universitas Padjadjaran (Other); Health Development Policy Agency, Ministry of Health Republic of Indonesia (Unknown); Coalition for Epidemic Preparedness Innovations (Other); The Peter Doherty Institute for Infection and Immunity (Other); Indonesia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RCH HREC Ref 81803
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
Keywords: Booster; fractional and standard doses; Pfizer; Astrazeneca; Moderna; COVID-19 vaccination; mRNA vaccine
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; ChAdOx1 nCoV-19; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A unblinded vaccinator will administer the dose and will not be involved in outcome assessment. Unblinding will occur for each participant at approximately 28 days after the study vaccine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- Pfizer-BioNTech Standard dose after CoronaVac priming (Experimental): Pfizer-BioNTech (BNT162b2, or Comirnaty®) Dose: 30ug in 0.3ml
  The 50 participants in this arm received second CoronaVac priming dose at least 6 months prior to randomisation.
  Interventions: Biological: Pfizer-BioNTech Standard dose
- Pfizer-BioNTech Fractional dose after CoronaVac priming (Experimental): Pfizer-BioNTech (BNT162b2, or Comirnaty®) Dose: 15ug in 0.15ml
  The 50 participants in this arm received second CoronaVac priming dose at least 6 months prior to randomisation.
  Interventions: Biological: Pfizer-BioNTech Fractional dose
- AstraZeneca Standard dose after CoronaVac priming (Experimental): AstraZeneca (ChAdOx1-S, Vaxzevria®). Dose: 0.5ml
  The 50 participants in this arm received second CoronaVac priming dose at least 6 months prior to randomisation.
  Interventions: Biological: AstraZeneca Standard dose
- AstraZeneca Fractional dose after CoronaVac priming (Experimental): AstraZeneca (ChAdOx1-S, Vaxzevria®). Dose: 0.25ml
  The 50 participants in this arm received second CoronaVac priming dose at least 6 months prior to randomisation.
  Interventions: Biological: AstraZeneca Fractional dose
- Moderna Standard Dose after CoronaVac priming (Experimental): Moderna (mRNA-1273 or Spikevax®) Dose: 50ug in 0.25ml
  The 100 participants in this arm received second CoronaVac priming dose at least 6 months prior to randomisation.
  Interventions: Biological: Moderna Standard dose
- Moderna Fractional Dose after CoronaVac priming (Experimental): Moderna (mRNA-1273 or Spikevax®) Dose: 20ug in 0.1ml
  The 100 participants in this arm received second CoronaVac priming dose at least 6 months prior to randomisation.
  Interventions: Biological: Moderna Fractional dose
- Pfizer-BioNTech Standard dose after AstraZeneca priming (Experimental): Pfizer-BioNTech (BNT162b2, or Comirnaty®) Dose: 30ug in 0.3ml
  The 50 participants in this arm received second AstraZeneca priming dose at least 6 months prior to randomisation.
  Interventions: Biological: Pfizer-BioNTech Standard dose
- Pfizer-BioNTech Fractional dose after AstraZeneca priming (Experimental): Pfizer-BioNTech (BNT162b2, or Comirnaty®) Dose: 15ug in 0.15ml
  The 50 participants in this arm received second AstraZeneca priming dose at least 6 months prior to randomisation.
  Interventions: Biological: Pfizer-BioNTech Fractional dose
- AstraZeneca Standard dose after AstraZeneca priming (Experimental): AstraZeneca (ChAdOx1-S, Vaxzevria®). Dose: 0.5ml
  The 50 participants in this arm received second AstraZeneca priming dose at least 6 months prior to randomisation.
  Interventions: Biological: AstraZeneca Standard dose
- AstraZeneca Fractional dose after AstraZeneca priming (Experimental): AstraZeneca (ChAdOx1-S, Vaxzevria®). Dose: 0.25ml
  The 50 participants in this arm received second AstraZeneca priming dose at least 6 months prior to randomisation.
  Interventions: Biological: AstraZeneca Fractional dose
- Moderna Standard Dose after AstraZeneca priming (Experimental): Moderna (mRNA-1273 or Spikevax®) Dose: 50ug in 0.25ml
  The 100 participants in this arm received second AstraZeneca priming dose at least 6 months prior to randomisation.
  Interventions: Biological: Moderna Standard dose
- Moderna Fractional Dose afterAstraZeneca priming (Experimental): Moderna (mRNA-1273 or Spikevax®) Dose: 20ug in 0.1
  The 100 participants in this arm received second AstraZeneca priming dose at least 6 months prior to randomisation.
  Interventions: Biological: Moderna Fractional dose

INTERVENTIONS:
Biological: Pfizer-BioNTech Standard dose — Standard Dose - (30ug in 0.3ml)
  The Pfizer-BioNTech COVID-19 vaccine, BNT162b2, encodes a P2 mutant spike protein and is formulated as an RNA-lipid nanoparticle (LNP) of nucleoside-modified mRNA (modRNA).
  Other Names: BNT162b2; Comirnaty
  Arms: Pfizer-BioNTech Standard dose after AstraZeneca priming; Pfizer-BioNTech Standard dose after CoronaVac priming
Biological: AstraZeneca Standard dose — Standard Dose (5xE10vp in 0.5ml)
  ChAdOx1 nCoV-19 is a recombinant replication-defective chimpanzee adenovirus expressing the SARS-CoV-2 spike (S) surface glycoprotein
  Other Names: ChAdOx1-S; Vaxzevria
  Arms: AstraZeneca Standard dose after AstraZeneca priming; AstraZeneca Standard dose after CoronaVac priming
Biological: Pfizer-BioNTech Fractional dose — Fractional Dose - (15ug in 0.15ml)
  The Pfizer-BioNTech COVID-19 vaccine, BNT162b2, encodes a P2 mutant spike protein and is formulated as an RNA-lipid nanoparticle (LNP) of nucleoside-modified mRNA (modRNA).
  Other Names: BNT162b2; Comirnaty
  Arms: Pfizer-BioNTech Fractional dose after AstraZeneca priming; Pfizer-BioNTech Fractional dose after CoronaVac priming
Biological: AstraZeneca Fractional dose — Fractional Dose (2.5E10vp in 0.25ml)
  ChAdOx1 nCoV-19 is a recombinant replication-defective chimpanzee adenovirus expressing the SARS-CoV-2 spike (S) surface glycoprotein
  Other Names: ChAdOx1-S; Vaxzevria
  Arms: AstraZeneca Fractional dose after AstraZeneca priming; AstraZeneca Fractional dose after CoronaVac priming
Biological: Moderna Standard dose — Standard dose (50ug in 0.25ml)
  Other Names: mRNA-1273; Spikevax®
  Arms: Moderna Standard Dose after AstraZeneca priming; Moderna Standard Dose after CoronaVac priming
Biological: Moderna Fractional dose — Fractional dose (20ug in 0.1ml)
  Other Names: mRNA-1273; Spikevax®
  Arms: Moderna Fractional Dose after CoronaVac priming; Moderna Fractional Dose afterAstraZeneca priming

SUMMARY:
This is a randomised controlled clinical trial to determine the reactogenicity and immunogenicity of booster doses of SARS-CoV-2 vaccines (Pfizer-BioNTech, AstraZeneca or Moderna) in adults who have previously received either AstraZeneca or Coronavac as their primary doses.

Both fractional and standard doses of Pfizer-BioNTech, AstraZeneca and Moderna will be tested.

DETAILED DESCRIPTION:
There will be a total of 800 participants in the study, to be randomised and administered booster doses in this study.

The study will be conducted at 3 clinics in Bandung. Participants will have previously received primary doses of Coronavac or Astranzeneca, with the second dose administered at least 6 months previously.

Participants will be followed for 12 months following the booster vaccine adminstration, with blood samples drawn at baseline, 28 days, 6 months and 12 months following booster vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy adults aged 18 years and above who had completed the primary series of COVID-19 vaccine with CoronaVac or AstraZeneca more than 6 months prior to enrolment to the study.
2. Signed written informed consent form and willing to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Those who have already received a third dose of SARS-CoV-2 vaccine
2. Concomitantly enrolled or scheduled to be enrolled in another trial.
3. Those with fever (temperature ˃ 37.5℃, measured with infrared thermometer/thermal gun), upper respiratory tract infection symptoms such as sneezing, nasal congestion, runny nose, cough, sore throat, loss of taste, chills and shortness of breath within 72 hours before enrolment.
4. Blood pressure ˃ 180/110 mmHg.
5. History of confirmed COVID-19 within one month prior to study enrolment.
6. History of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnoea, and angioneurotic oedema.
7. Those with uncontrolled autoimmune disease such as systemic lupus erythematosis.
8. History of uncontrolled coagulopathy or blood disorders, immune deficiency.
9. History of having received blood derived product/transfusion within 3 months prior to enrolment.
10. Those who received immunosuppressant therapy such as high-dose corticosteroid or cancer chemotherapy
11. Those with uncontrolled chronic disease, such as severe heart disease, asthma exacerbation
12. Those who have history of uncontrolled epilepsy (within the last 2 years) or other progressive neurological disorders, such as Guillain-Barre Syndrome
13. Those who have receive any vaccination within 2 weeks before study vaccine administration for this protocol, or intended to receive any vaccination within 2 weeks after study vaccine administration.
14. Pregnant woman
15. Those aged ≥60 years old with difficulty in climbing 10 steps of stairs, frequently experiencing fatigue, difficulty in walking 100-200 m, or having at least 5 comorbidities (hypertension, diabetes, cancer, chronic lung disease, heart attack, congestive heart failure, chest pain, asthma, joint pain, stroke, and kidney disease).
16. Those who are study staff working on the study or the immediate family of study investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 specific Immunoglobulin (Ig)G antibodies at 28-days post booster vaccination | Assessed at 28 days
  Serum samples collected at 28-days post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using IgG CMIA. The primary endpoint is the seroresponse rate at the Day-28 visit. The Seroresponse rate at the individual level is defined as either a ≥4-fold rise in binding antibodies at the Day-28 visit compared to baseline (pre-vaccination) with a titre of <200 BAU/ml, a ≥2-fold rise among participants with a baseline (pre-vaccination) titre of >≥200 BAU/ml, or ≥4 times the lower limit of detection if baseline levels are lower than the limit of detection.
Incidence of solicited systemic and local reactions (reactogenicity) | Assessed for 7 days post-vaccination
  Questionnaire to document solicited reactions is developed specifically for this study. Data will be reported as the proportion of participants who report grade 3 or 4 reactions by each intervention arm. Solicited reactions such as pain, tenderness, erythema/redness, induration, swelling, fever, nausea, vomiting, headache, fatigue/malaise, myalgia, arthralgia, diarrhea, enlarged lymph nodes will be collected from the participants 7 days post-vaccination.

SECONDARY OUTCOMES:
SARS-CoV-2 specific IgG antibodies at baseline (pre booster), 6- and 12-months post booster vaccination. | Assessed at time-points: baseline, 28 days, 6 months, and 12 months).
  Serum samples collected at baseline (pre booster), 28 days, and 6- and 12-months post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using IgG CMIA. Data will be reported as binding antibody units (BAU)/mL and presented as geometric mean concentration (GMC) and 95% confidence intervals (CI)
SARS-CoV-2 specific neutralising antibodies at baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination measured by surrogate virus neutralization test (sVNT) | Assessed at 4 time-points (baseline, 28 days, 6 months, and 12 months).
  Serum samples collected at baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific neutralising antibodies using the GenScript® cPass surrogate virus neutralization test (sVNT) for both wild-type and Omicron variant. Neutralising antibody response will be reported as percentage (%) inhibition of receptor binding domain-angiotensin-converting enzyme 2 (RBD-ACE2) binding relative to a positive control.
SARS-CoV-2 specific neutralising antibodies at baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination measured by SARS-CoV-2 microneutralisation assay | Assessed at 4 time-points (baseline, 28 days, 6 months, and 12 months).
  A subset of samples from all four timepoints will be assessed using a SARS-CoV-2 microneutralisation assay to both the wild type (vaccine) strain and for two SARS-CoV-2 Variants of concern. Neutralizing antibody will be reported as endpoint titre.
Interferon gamma (IFNγ) concentrations in International Units (IU)/mL | Assessed at 4 time-points (baseline, 28 days, 6 months, and 12 months).
  Applicable to the subset participants with additional blood collection. Interferon gamma (IFNγ) concentrations as a measurement of cellular immunity will be assessed on a subset of the participants from each group. QuantiFERON Human IFN-γ SARS-CoV-2 (Qiagen) will be used to stimulate IFN-γ production in peripheral blood mononuclear cells (PBMCs) and then IFN-γ production will be measured using ELISA (enzyme-linked immunosorbent assay). Data will be presented as geometric mean concentration (GMC) and 95% confidence intervals (CI).
Number of IFNγ producing cells/million PBMCs | Assessed at 4 time-points (baseline, 28 days, 6 months, and 12 months).
  Applicable to the subset participants with additional blood collection. IFNγ producing cells as a measurement of cellular immunity will be assessed on a subset of the participants from each group. IFN-γ Enzyme-Linked ImmunoSpot (Elispot) assay will be performed on isolated peripheral blood mononuclear cells (PBMCs). Data will be reported as number of IFNγ producing cells/million and presented using means and 95% confidence intervals.
Frequency of cytokine-expressing T cells | Assessed at 4 time-points (baseline, 28 days, 6 months, and 12 months).
  Applicable to the subset participants with additional blood collection. Frequency of cytokine-expressing T cells will be assessed on a subset of participants using Flow cytometry (intracellular staining) on PBMCs samples. Data will be reported as frequency (%) of cytokine-expressing T cells presented as means and 95% CI.
Cytokine concentrations following PBMCs stimulation | Assessed at 4 time-points (baseline, 28 days, 6 months, and 12 months).
  Applicable to the subset participants with additional blood collection. Cytokine concentrations following PBMCs stimulation will be assessed on a subset (40%) of participants using multiplex cytokine assays.Data will be reported as cytokine concentrations in pg/ml and presented as GMC and 95% CI.IFN-γ Elispot, intracellular cytokine assays (flow cytometry) and multiplex cytokine assays will be performed on isolated peripheral blood mononuclear cells (PBMCs)
Incidence of unsolicited adverse events (AE) | 28 days post booster vaccination for all AE
  All unsolicited AE will be collected for 28 days post booster vaccination. Data will be presented as proportion of participants who report unsolicited AE.
Incidence of medically attended adverse events | 3 months post booster vaccination for medically attended AE
  Participants with medically attended AE will be collected for 3 months post booster vaccination. Data will be presented as proportion of participants who report unsolicited AE
Incidence of serious adverse events (SAE) | 12 months post booster vaccination for SAE
  SAE will be collected throughout the follow up period of 12 months. Data will be presented as a proportion of participants who report SAE.
Incidence of confirmed COVID-19 infection | Throughout the follow up period of 12 months.
  Confirmed (Polymerase Chain Reaction [PCR] or rapid antigen test) COVID-19 infections will be documented throughout the follow-up period, by clinical severity

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Fadlyana, Dr, Principal Investigator — Universitas Padjadjaran, Indonesia
Locations (3):
- Indonesia (3):
  - Puskesmas Ciumbuleuit, Bandung, West Java
  - Puskesmas Dago, Bandung, West Java
  - Puskesmas Garuda, Bandung, West Java

IPD SHARING:
Plan to Share IPD: Yes
We will share data to ethically approved studies in cases where participants have indicated on consent form that they consent to this use of their data and where consistent with terms of collaboration agreement/s
Supporting Information: Study Protocol, ICF
Time Frame: IPD sharing plans in development
Access Criteria: IPD sharing plans in development